CLINICAL TRIAL: NCT02118714
Title: A Multicenter, Single-Arm Study of the Effects of Atrasentan on Spermatogenesis and Testicular Function
Brief Title: Atrasentan Spermatogenesis and Testicular Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M12-919; 2016-000722-19 (EudraCT Number)
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Nephropathy; Diabetes
Keywords: Diabetic Nephropathies; Kidney Diseases; Urologic Diseases; Diabetes Complications; Diabetes Mellitus; Endocrine System Diseases
MeSH Terms: conditions — Kidney Diseases; Diabetes Mellitus; Diabetic Nephropathies; Urologic Diseases; Diabetes Complications; Endocrine System Diseases | interventions — Atrasentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atrasentan (Experimental): Atrasentan 0.75 mg administered orally once daily (QD) for 26 weeks
  Interventions: Drug: Atrasentan

INTERVENTIONS:
Drug: Atrasentan — Atrasentan

SUMMARY:
This study is being conducted to evaluate the effects of Atrasentan on sperm production and testicular function in male subjects with Type 1 or 2 Diabetes and Nephropathy.

This study included 2 periods: a Treatment Period (up to 26 weeks) followed by an Observational Period (up to an additional 52 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Males 30 to 75 years of age
* Type 1 or 2 diabetes and receiving treatment with at least one anti-hyperglycemic medication and angiotensin-converting enzyme inhibitors (ACEi)/angiotensin receptor blockers (ARB) (renin-angiotensin system [RAS] inhibitor)
* Estimated Glomerular Filtration Rate (eGFR) equal to or greater than 35 mL/min/1.73 m^2 with the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Formula and Urine Albumin-to-Creatinine Ratio (UACR) equal to or greater than 30 and less than 5,000 mg/g creatinine.
* Able to provide a semen specimen at the required intervals.
* Baseline sperm concentration equal to or greater than 30 million per mL.

Exclusion Criteria:

* Treatment with hormone suppressive agents or cancer chemotherapy within the 6 months prior to the initial screening visit or planned during the study.
* History of severe peripheral edema or facial edema unrelated to trauma or history of myxedema in the prior 4 weeks prior to screening.
* History of pulmonary hypertension, pulmonary fibrosis or any lung disease requiring oxygen therapy.
* Documented diagnosis of heart failure, previous hospitalization for heart failure or current or constellation of symptoms (dyspnea on exertion, pedal edema, orthopnea, paroxysmal nocturnal dyspnea) felt to be compatible with heart failure, that was not explained by other causes, and for which there was a change in medication or other management directed at heart failure.
* Currently receiving or has received hormone replacement therapy within 6 months prior to screening.

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04-06 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (13):
- United States (9):
  - Alliance Research Centers /ID# 125945, Laguna Hills, California
  - Frank Clark Urology Center /ID# 147794, Santa Monica, California
  - Research by Design, LLC /ID# 160784, Evergreen Park, Illinois
  - Southern IL Univ School of Med /ID# 129010, Springfield, Illinois
  - Crescent City Clinical Res Ctr /ID# 150989, Metairie, Louisiana
  - Tulane Univ /ID# 130308, New Orleans, Louisiana
  - Albany Medical College /ID# 131068, Albany, New York
  - Urologic Consultants of Southeastern Pennsylvania /ID# 124277, Bala-Cynwyd, Pennsylvania
  - Eastern Virginia Med School /ID# 153740, Norfolk, Virginia
- Charite Research Organisation GmbH /ID# 154264, Berlin, Germany
- Italy (2):
  - Ospedale S. Carlo Borromeo /ID# 151672, Milan
  - SCDU Nefrologia e dialisi-CMID /ID# 151673, Torino
- Hospital Universitario Reina S /ID# 151692, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: http://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Safety Analysis Set included all enrolled participants who received >= 1 dose of Atrasentan (N = 20); of these 20, 6 participants entered an Observational Period of up to an additional 52 weeks.
Groups:
- Atrasentan: Atrasentan 0.75 mg administered orally once daily (QD).
Period: Overall Study
Arm/Group | Atrasentan
Started | 20
Completed | 17
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Arm/Group | Atrasentan
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a Sperm Concentration < 15 Million Per mL by Treatment Week 26
Description: Percentage of Subjects with a Sperm Concentration < 15 million per mL by Treatment Week 26. Sperm concentration was calculated as measure of the number sperm per milliliter of semen. Duplicate semen samples were collected. The average of the 2 samples were used as the value for that scheduled collection period.
Time Frame: Up to 26 weeks
Population: Evaluable Set: Subjects who met 1 of the following: Study drug compliance ≥ 70%, completed Treatment Period, all planned sperm samples collected; or 2) at least 1 dose study drug, a sperm concentration value that was <15 million/mL observed by the end of the Treatment Period or had a ≥50% reduction from Baseline at the end of the Treatment Period.
Measure: Number; unit: percentage of participants
Arm/Group | Atrasentan
Number analyzed (Participants) | 17
percentage of participants | 23.5
Statistical Analysis 1: Comparison: Atrasentan; Test type: Other; Percentage of Participants = 23.5, 80% CI 2-sided [10.7 to 41.6]
Statistical Analysis 2: Comparison: Atrasentan; Test type: Other; Percentage of Participants = 23.5, 95% CI 2-sided [6.8 to 49.9]

2. Secondary Outcome: Percentage of Participants Who Entered the Observation Period and Did Not Return to Within 15% of Baseline Sperm Concentration or Above During the 52-Week Observational Period
Description: The percentage of participants who entered the Observational Period and did not return to within 15% of Baseline sperm concentration or above during the 52-week Observational Period. Duplicate semen samples were to be collected during the Observational Period. Sperm concentration was calculated as measure of the number sperm per milliliter of semen. Duplicate semen samples were collected. The average of the 2 samples were used as the value for that scheduled collection period.
Time Frame: Up to 52 weeks after the Treatment Period
Population: Evaluable Set
Measure: Number; unit: percentage of participants
Arm/Group | Atrasentan
Number analyzed (Participants) | 17
percentage of participants | 11.8
Statistical Analysis 1: Comparison: Atrasentan; Test type: Other; Percentage of Participants = 11.8, 80% CI 2-sided [3.2 to 28.4]
Statistical Analysis 2: Comparison: Atrasentan; Test type: Other; Percentage of Participants = 11.8, 95% CI 2-sided [1.5 to 36.4]

3. Secondary Outcome: Change From Baseline up to Treatment Period Week 26 and Observation Period Week 52 in Sperm Concentration
Description: Duplicate semen samples will be collected during the Treatment and Observational Periods. The average of the 2 samples were used as the value for that scheduled collection period. A negative change from baseline indicated a decrease in sperm concentration.
Time Frame: From Week 0 up to Treatment Period Week 26 and Observation Period Week 52
Population: All participants in the Safety Analysis Set (defined as enrolled participants who receive >= 1 dose of Atrasentan) with evaluable data at both baseline and the given time point.
Measure: Mean (Standard Deviation); unit: sperm * million per milliliter(X10^6/mL)
Arm/Group | Atrasentan
Number analyzed (Participants) | 18
sperm * million per milliliter(X10^6/mL)
  Treatment Period Week 13 | 2.2 (42.21)
  Treatment Period Week 26: number analyzed (Participants) | 17
  Treatment Period Week 26 | -10.6 (53.44)
  Observation Period Week 13: number analyzed (Participants) | 6
  Observation Period Week 13 | 35.8 (113.60)
  Observation Period Week 26: number analyzed (Participants) | 2
  Observation Period Week 26 | -16.5 (0.00)
  Observation Period Week 39: number analyzed (Participants) | 2
  Observation Period Week 39 | -27.5 (19.09)
  Observation Period Week 52: number analyzed (Participants) | 2
  Observation Period Week 52 | -25.8 (1.06)

4. Secondary Outcome: Change From Baseline up to Treatment Period Week 26 and Observation Period Week 52 in Sperm Motility
Description: Duplicate semen samples will be collected during the Treatment and Observation Periods. The average of the 2 samples were used as the value for that scheduled collection period. A negative change from baseline indicated a lower sperm motility (worsening).
Time Frame: From Week 0 up to Treatment Period Week 26 and Observation Observation Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent motility
Arm/Group | Atrasentan
Number analyzed (Participants) | 18
percent motility
  Treatment Period Week 13 | -5.8 (13.65)
  Treatment Period Week 26: number analyzed (Participants) | 17
  Treatment Period Week 26 | -7.4 (15.77)
  Observation Period Week 13: number analyzed (Participants) | 6
  Observation Period Week 13 | -0.3 (19.20)
  Observation Period Week 26: number analyzed (Participants) | 2
  Observation Period Week 26 | -6.3 (5.30)
  Observation Period Week 39: number analyzed (Participants) | 2
  Observation Period Week 39 | 10.8 (15.20)
  Observation Period Week 52: number analyzed (Participants) | 2
  Observation Period Week 52 | 1.8 (16.62)

5. Secondary Outcome: Change From Baseline up to Treatment Period Week 26 and Observation Period Week 52 in Sperm Morphology
Description: Duplicate semen samples will be collected during the Treatment and Observational Periods. The percentage of sperm with normal versus abnormal morphology will be determined via microscopic analysis. A positive change from baseline indicates an improved sperm morphology.
Time Frame: From Week 0 up to Treatment Period Week 26 and Observation Period Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of normal
Arm/Group | Atrasentan
Number analyzed (Participants) | 18
percentage of normal
  Treatment Period Week 13 | -1.1 (4.78)
  Treatment Period Week 26: number analyzed (Participants) | 17
  Treatment Period Week 26 | -2.2 (7.54)
  Observation Period Week 13: number analyzed (Participants) | 6
  Observation Period Week 13 | -0.8 (7.53)
  Observation Period Week 26: number analyzed (Participants) | 2
  Observation Period Week 26 | -6.8 (0.35)
  Observation Period Week 39: number analyzed (Participants) | 2
  Observation Period Week 39 | -2.3 (1.77)
  Observation Period Week 52: number analyzed (Participants) | 2
  Observation Period Week 52 | 1.8 (0.35)

6. Secondary Outcome: Change From Baseline up to Treatment Period Week 26 and Observation Period Week 52 in Semen Volume
Description: Duplicate semen samples will be collected during the Treatment and Observation Periods. The average of the 2 samples were used as the value for that scheduled collection period. A negative change from baseline indicated a decrease in semen volume.
Time Frame: From Week 0 to up to Treatment Period Week 26 and Observation Period Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Atrasentan
Number analyzed (Participants) | 18
milliliter (mL)
  Treatment Period Week 13 | 0.0 (0.65)
  Treatment Period Week 26: number analyzed (Participants) | 17
  Treatment Period Week 26 | -0.3 (0.75)
  Observation Period Week 13: number analyzed (Participants) | 6
  Observation Period Week 13 | 0.0 (1.39)
  Observation Period Week 26: number analyzed (Participants) | 2
  Observation Period Week 26 | 0.0 (0.35)
  Observation Period Week 39: number analyzed (Participants) | 2
  Observation Period Week 39 | 0.1 (0.42)
  Observation Period Week 52: number analyzed (Participants) | 2
  Observation Period Week 52 | -0.4 (0.14)

7. Secondary Outcome: Change From Baseline up to Treatment Period Week 26 and Observation Period Week 52 in Serum Testosterone
Description: Serum hormones levels will be tested during the Treatment and Observational Periods. A negative change from baseline indicated a decrease in serum testosterone.
Time Frame: From Week 0 up to Treatment Period Week 26 and Observation Period Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanomole/liter (nmol/L)
Arm/Group | Atrasentan
Number analyzed (Participants) | 18
nanomole/liter (nmol/L)
  Treatment Period Week 13 | 0.2 (2.18)
  Treatment Period Week 26 | 0.8 (2.33)
  Observation Period Week 13: number analyzed (Participants) | 5
  Observation Period Week 13 | 0.6 (2.08)
  Observation Period Week 26: number analyzed (Participants) | 3
  Observation Period Week 26 | -0.3 (0.85)
  Observation Period Week 39: number analyzed (Participants) | 2
  Observation Period Week 39 | -1.6 (1.37)
  Observation Period Week 52: number analyzed (Participants) | 2
  Observation Period Week 52 | -1.1 (1.68)

8. Secondary Outcome: Change From Baseline up to Treatment Period Week 26 and Observation Period Week 52 in Estradiol
Description: Serum hormones levels were tested during the Treatment and Observational Periods. A negative change from baseline indicated a decrease in serum estradiol.
Time Frame: From Week 0 up to Treatment Period Week 26 and Observation Period Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Picomoles Per Litre (pmol/L)
Arm/Group | Atrasentan
Number analyzed (Participants) | 18
Picomoles Per Litre (pmol/L)
  Treatment Period Week 13 | -11.7 (44.57)
  Treatment Period Week 26 | -18.6 (42.04)
  Observation Period Week 13: number analyzed (Participants) | 6
  Observation Period Week 13 | -17.8 (62.78)
  Observation Period Week 26: number analyzed (Participants) | 3
  Observation Period Week 26 | -47.3 (39.97)
  Observation Period Week 39: number analyzed (Participants) | 2
  Observation Period Week 39 | 20.3 (4.78)
  Observation Period Week 52: number analyzed (Participants) | 2
  Observation Period Week 52 | 10.5 (45.54)

9. Secondary Outcome: Change From Baseline up to Treatment Period Week 26 and Observation Period Week 52 in Lutenizing Hormone (LH)
Description: Serum hormones levels will be tested during the Treatment and Observational Periods. A positive change from baseline indicated an increase in serum lutenizing hormone.
Time Frame: From Week 0 to up to Treatment Period Week 26 and Observation Period Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International Units/Liter (IU/L)
Arm/Group | Atrasentan
Number analyzed (Participants) | 18
International Units/Liter (IU/L)
  Treatment Period Week 13 | 1.0 (2.60)
  Treatment Period Week 26 | 0.7 (2.44)
  Observation Period Week 13: number analyzed (Participants) | 6
  Observation Period Week 13 | 1.3 (1.33)
  Observation Period Week 26: number analyzed (Participants) | 3
  Observation Period Week 26 | 1.9 (2.35)
  Observation Period Week 39: number analyzed (Participants) | 2
  Observation Period Week 39 | 0.5 (0.07)
  Observation Period Week 52: number analyzed (Participants) | 2
  Observation Period Week 52 | 1.8 (3.46)

10. Secondary Outcome: Change From Baseline up to Treatment Period Week 26 and Observation Period Week 52 in in Follicle Stimulating Hormone (FSH)
Description: Serum hormones levels will be tested during the Treatment and Observational Periods. A positive change from baseline indicated an increase in serum follicle stimulating hormone.
Time Frame: From Week 0 to Treatment Week 26 and Observation Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International Units/Liter (IU/L)
Arm/Group | Atrasentan
Number analyzed (Participants) | 18
International Units/Liter (IU/L)
  Treatment Period Week 13 | 1.1 (2.43)
  Treatment Period Week 26 | 0.8 (1.91)
  Observation Period Week 13: number analyzed (Participants) | 6
  Observation Period Week 13 | 0.4 (1.60)
  Observation Period Week 26: number analyzed (Participants) | 3
  Observation Period Week 26 | 0.7 (1.49)
  Observation Period Week 39: number analyzed (Participants) | 2
  Observation Period Week 39 | 0.4 (1.57)
  Observation Period Week 52: number analyzed (Participants) | 2
  Observation Period Week 52 | 0.8 (0.59)

11. Secondary Outcome: Change From Baseline up to Treatment Period Week 26 and Observation Period Week 52 in Inhibin B
Description: Serum hormones levels will be tested during the Treatment and Observational Periods. A negative change from baseline indicated a decrease in serum Inhibin B.
Time Frame: From Week 0 up to Treatment Period Week 26 and Observation Period Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Atrasentan
Number analyzed (Participants) | 18
picogram per milliliter (pg/mL)
  Treatment Period Week 13 | -2.7 (24.19)
  Treatment Period Week 26 | -8.8 (34.73)
  Observation Period Week 13: number analyzed (Participants) | 6
  Observation Period Week 13 | -7.2 (20.77)
  Observation Period Week 26: number analyzed (Participants) | 3
  Observation Period Week 26 | -22.7 (27.10)
  Observation Period Week 39: number analyzed (Participants) | 2
  Observation Period Week 39 | -21.0 (16.97)
  Observation Period Week 52: number analyzed (Participants) | 2
  Observation Period Week 52 | -5.5 (2.12)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to approximately 30 weeks).
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening reported by a participant from the time that the first dose of atrasentan is administered until 30 days have elapsed following discontinuation of adalimumab administration. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Atrasentan
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atrasentan (N=20)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
POSTOPERATIVE RESPIRATORY FAILURE (Injury, poisoning and procedural complications) | 1 (1)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 2 (3)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
AORTIC DISSECTION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atrasentan (N=20)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 1 (1)
LEFT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 1 (1)
EUSTACHIAN TUBE DYSFUNCTION (Ear and labyrinth disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (3)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
TOOTH DISORDER (Gastrointestinal disorders) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 4 (4)
BRONCHITIS (Infections and infestations) | 1 (1)
LOCALISED INFECTION (Infections and infestations) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 4 (5)
PNEUMONIA (Infections and infestations) | 1 (2)
TINEA CRURIS (Infections and infestations) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 1 (1)
CHEST INJURY (Injury, poisoning and procedural complications) | 1 (1)
POST PROCEDURAL INFLAMMATION (Injury, poisoning and procedural complications) | 1 (1)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1)
BLOOD PRESSURE INCREASED (Investigations) | 1 (1)
WEIGHT INCREASED (Investigations) | 1 (1)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 (1)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (2)
DELIRIUM TREMENS (Psychiatric disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
PANIC ATTACK (Psychiatric disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1)
POLLAKIURIA (Renal and urinary disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DENTAL PROSTHESIS USER (Social circumstances) | 1 (1)
AORTIC ANEURYSM (Vascular disorders) | 1 (1)
HAEMATOMA (Vascular disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1)
ORTHOSTATIC HYPERTENSION (Vascular disorders) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT02118714/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT02118714/SAP_001.pdf